CLINICAL TRIAL: NCT01523756
Title: An Open-labelled Randomized Cross-over and Controlled Exploratory Investigation Comparing Several Variants of a Newly Developed Ostomy Appliance With Regard to Performance in 20 Patients With Ileostomy
Brief Title: A Clinical Investigation of New Ostomy Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CP226
Record Dates: First submitted 2012-01-10; First posted 2012-02-01 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-01

CONDITIONS: Leakage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- test product 1 first (Experimental): own product (baseline) - test product 1 - test product 2
  test product 1 = New ostomy base plate. Due to company confidentiality the product is just called test product 1
  Interventions: Device: test product 1: new ostomy base plate with Coloplast as manufacturer
- test product 2 first (Experimental): own product (baseline) - test product 2 - test product 1
  test product 2 = New ostomy base plate. Due to company confidentiality the product is just called test product 2
  Interventions: Device: test product 2: new ostomy base plate with Coloplast as manufacturer

INTERVENTIONS:
Device: test product 1: new ostomy base plate with Coloplast as manufacturer — test product 1 is tested first
  Arms: test product 1 first
Device: test product 2: new ostomy base plate with Coloplast as manufacturer — test product 2 is tested first
  Arms: test product 2 first

SUMMARY:
This is an open-labelled randomized cross-over and controlled exploratory intervention that aims to include 20-30 patients with an ileostomy. Every patient is to test two new ostomy appliances each for two weeks. During the test a questionaire is to be filled out and interviews will take place. Primary parameter is leakage. A Study nurse will visit the participants in their homes every two week during the test.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Have had an ileostomy for more than 3 months.
3. Have used convex products for the last 1 month.
4. Has given written Informed Consent.
5. Have an ileostomy with a diameter between 15 and 33 mm.
6. Have inward peristomal area

Exclusion Criteria:

1. Have loop ostomy
2. Pregnant or breastfeeding.
3. Known allergy towards any of the product components or ingredients.
4. Currently receiving or have within the last 2 months received radio- and/or chemotherapy.
5. Currently receiving or have within the past month received local or systemic steroid treatment in the peristomal area.
6. Currently suffering from peristomal skin problems (i.e. bleeding or red and broken skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited through the Coloplast database.
Groups:
- Own Product (Baseline) - Test Product 1 - Test Product 2: own product (baseline) - test product 1 - test product 2
  test product 1 = New ostomy base plate. Due to company confidentiality the product is just called test product 1
- Own Product (Baseline) - Test Product 2 - Test Product 1: own product (baseline) - test product 2 - test product 1
  test product 2 = New ostomy base plate. Due to company confidentiality the product is just called test product 2
Period: Baseline Period
Arm/Group | Own Product (Baseline) - Test Product 1 - Test Product 2 | Own Product (Baseline) - Test Product 2 - Test Product 1
Started | 11 | 9
Completed | 11 | 8
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Test Period 1
Arm/Group | Own Product (Baseline) - Test Product 1 - Test Product 2 | Own Product (Baseline) - Test Product 2 - Test Product 1
Started | 11 | 8
Completed | 10 | 8
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Test Period 2
Arm/Group | Own Product (Baseline) - Test Product 1 - Test Product 2 | Own Product (Baseline) - Test Product 2 - Test Product 1
Started | 10 | 8
Completed | 10 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Leakage Under the Base Plate Using a 24-point Scale
Description: Leakage under the baseplate was measured with a 24 point scale where 0 points represents no leakage (best possible out come) and 24 points represents leakage on the whole plate (worst possible outcome)
Time Frame: Each product will be tested 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: degree of leakage on the baseplate
Groups:
- Test Product 1: own product (baseline) - test product 1 - test product 2
  test product 1 = New ostomy base plate. Due to company confidentiality the product is just called test product 1
- Test Product 2: own product (baseline) - test product 2 - test product 1
  test product 2 = New ostomy base plate. Due to company confidentiality the product is just called test product 2
- Baseline: Data collected on own product-
  All subjects collected baseline data on own product in the first period.
Arm/Group | Test Product 1 | Test Product 2 | Baseline
Number analyzed (Participants) | 19 | 18 | 20
Number analyzed (degree of leakage on the baseplate) | 111 | 111 | 113
units on a scale | 4.5 (5.3) | 3.3 (4.3) | 4.4 (4.7)

ADVERSE EVENTS:
Arm/Group | Test Product 1 | Test Product 2 | Baseline
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 8/19 | 6/18 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product 1 (N=20) | Test Product 2 (N=20) | Baseline (N=20)
Gastroenterit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product 1 (N=19) | Test Product 2 (N=18) | Baseline (N=20)
Skin irritation (peristomal) (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Bleeding peristomal skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Itchy peristomal skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Gastroenterit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to the testproducts
Urin retension (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to the testproducts
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) — Not related to the testproducts
febrilia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Not related to the testproducts
pain in bladder/Tenesmi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to the testproducts
Nausea (General disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to the testproducts
elevated prostataspecific antigen (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to the testproducts
skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to the testproducts
cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) — Not related to the testproducts
sclerose attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to the testproducts
Herpes on the back of the thigh (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to the testproducts
candidiacis on labia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — candidadiacis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes